CLINICAL TRIAL: NCT05420441
Title: Chitosan Versus Glucosamine Phonophoresis in the Management of Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: Chitosan Versus Glucosamine Phonophoresis in the Management of Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy Ali Hassan ElMeligie, Principal investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChPhono2022
Record Dates: First submitted 2022-06-12; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Knee Osteoarthritis; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Phonophoresis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Phonophoresis with chitosan group) (Experimental): Patients in this group will receive chitosan through phonophoresis plus conventional treatment. For the phonophoresis parameters: pulsed ultrasonic waves (25%) of 1 MHz frequency and 1 W/cm2 intensity applied with a 5 cm diameter transducer. The total time of ultrasound application was eight minutes.Patients will also receive conventional Physical therapy program
  Interventions: Device: Phonophoresis with chitosan; Procedure: Conventional Physical Therapy
- Group B (Phonophoresis with glucosamine group) (Experimental): Patients in this group will receive glucosamine through phonophoresis plus conventional treatment. For the phonophoresis parameters: pulsed ultrasonic waves (25%) of 1 MHz frequency and 1 W/cm2 intensity applied with a 5 cm diameter transducer. The total time of ultrasound application was eight minutes.Patients will also receive conventional Physical therapy program.
  Interventions: Device: Phonophoresis with glucoasmine; Procedure: Conventional Physical Therapy
- Group C (Conventional physical therapy only) (Active Comparator): Patients in the control group will receive the conventional treatment for knee osteoarthritis only, which will include the application of TENS, pulsed ultrasound, infrared light and exercise.
  Interventions: Procedure: Conventional Physical Therapy

INTERVENTIONS:
Device: Phonophoresis with chitosan — Patients in this group will receive chitosan through phonophoresis plus conventional treatment. For the phonophoresis parameters: pulsed ultrasonic waves (25%) of 1 MHz frequency and 1 W/cm2 intensity applied with a 5 cm diameter transducer. The total time of ultrasound application was eight minutes.Patients will also receive conventional Physical therapy program
  Arms: Group A (Phonophoresis with chitosan group)
Device: Phonophoresis with glucoasmine — Patients in this group will receive glucosamine through phonophoresis plus conventional treatment. For the phonophoresis parameters: pulsed ultrasonic waves (25%) of 1 MHz frequency and 1 W/cm2 intensity applied with a 5 cm diameter transducer. The total time of ultrasound application was eight minutes.Patients will also receive conventional Physical therapy program.
  Arms: Group B (Phonophoresis with glucosamine group)
Procedure: Conventional Physical Therapy — Patients in the control group will receive the conventional treatment for knee osteoarthritis only, which will include the application of TENS, pulsed ultrasound, infrared light and exercise.

SUMMARY:
The study will be conducted to answer the following questions:

* Is there an effect of phonophoresis using glucosamine on pain level , function and range of motion in knee osteoarthritis patients ?
* Is there an effect of phonophoresis using chitosan on pain level , function and range of motion in knee osteoarthritis patients ?
* Is there a difference between the effect of phonophoresis using glucosamine and phonophoresis using chitosan on pain level , function and range of motion in knee osteoarthritis patients ?

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral grade II knee osteoarthritis (clinical and imaging diagnosis X-ray).
* knee pain intensity ≥ 5 on the Visual Analogue Scale (VAS)

Exclusion Criteria:

* Anterior Cruciate Ligament (ACL) and meniscus injury
* use of oral or injected corticosteroids in the last 3 months
* history of knee surgery or fracture
* acute infectious synovitis or arthritis conditions
* presence of malignancy
* individuals with, topical lesions, contact dermatitis and history of cutaneous hypersensitivity

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale | Baseline and Change from baseline pain scores at four weeks
  The visual analog scale (VAS) is a pain rating scale first used by Hayes and Patterson in 1921. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
Change in WOMAC INDEX | Baseline and Change from baseline scores at four weeks
  The WOMAC VA 3.1 Index score (WOMAC INDEX) is the sum of WOMAC A (total pain), WOMAC B (stiffness) and WOMAC C (functional impairment) subscores. The WOMAC INDEX score ranges from 0 to 2400 mm, with higher scores indicating higher disease burden.
Range of Motion at knee joint both in extension and flexion | Baseline and Change from baseline scores at four weeks
  The ROM will be measured using the Baseline 12-1056 bubble inclinometer. Patients will be in prone position and will be instructed to move their leg away from the thigh to measure extension range of motion and move the leg toward the thigh to measure flexion

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H ElGendy, Ph.D, Study Chair — Cairo University
Locations (1):
- El-Kasr El-Ainy hospital, Al Manyal, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No